CLINICAL TRIAL: NCT01153360
Title: Peri-operative Oral Triiodothyronine Replacement Therapy to Decrease the Risk of Transient Atrial Fibrillation After Off-pump Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Yong-Sun Choi, assistant professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2010-0086
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Non-thyroidal Illness Syndrome
MeSH Terms: conditions — Euthyroid Sick Syndromes | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T3 (Experimental): triiodothyronine
  Interventions: Drug: liothyronine sodium
- cyanocobalamin (Active Comparator): vitamin B12
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liothyronine sodium — liothyronine sodium 20ug, every 12hour (before anesthetic induction, total 4 times)
  Arms: T3
Drug: placebo — vitamin B12
  Arms: cyanocobalamin

SUMMARY:
This study is planned to medicate oral T3(Liothyronine)to the patients who are planned to have OPCAB(off- pump coronary bypass graft surgery. The aim of this study was to assess the effects of oral triiodothyronine (T3) therapy on postoperative thyroid hormone concentrations, hemodynamic variables and outcomes in patients undergoing OPCAB in a randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing Off-pump coronary artery bypass graft

Exclusion Criteria:

* No normal sinus rhythm,
* History of thyroid disease
* Abnormal thyroid hormone
* Renal dysfunction
* Hepatic dysfunction
* LVEF <30%
* Recent MI
* Active infection 1~15

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
compare the serum T3 concentrations and the number of patients with serum T3 concentrations below the normal range between the groups | until 36 hours after surgery

SECONDARY OUTCOMES:
difference of hemodynamic performance and myocardial injury | during surgery and 36 hr after surgery
  difference of hemodynamic performance and myocardial injury between the groups

OTHER OUTCOMES:
major morbidity endpoints including acute renal failure, cardiovascular failure, stroke, mediastinitis, need for ventilator support for >48 h, and new onset atrial fibrillation | until discharge of hospital

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Sun Choi, MD, Ph.D, Principal Investigator — Anesthesiology & Pain Medicine, Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea